CLINICAL TRIAL: NCT00923923
Title: Stress Reactivity in Veterans Receiving Pharmacological Treatment for Post-traumatic Stress Disorder (PTSD) and Alcohol Dependence
Brief Title: Stress Reactivity in Veterans Receiving Pharmacological Treatment for PTSD and Alcohol Dependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HIC # 0806003974; HSS # ER0005
Record Dates: First submitted 2009-06-12; First posted 2009-06-18 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Post-traumatic Stress Disorder; Alcohol Dependence
Keywords: stress reactivity; PTSD; alcohol dependence; drinking; craving
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- levels of stress (Experimental)
  Interventions: Behavioral: stress

INTERVENTIONS:
Behavioral: stress — compare levels of stress

SUMMARY:
Method: This study is designed as an accompaniment to an already funded study - a 12-week treatment trial with prazosin for patients with PTSD and AD.

The study design will consist of III phases. In phase I, all subjects will participate in three laboratory sessions to determine their reactivity to stress. Stress reactivity will be measured using: traumatic experiences, stressful non-trauma experiences and neutral experiences, presented randomly. Laboratory sessions will be conducted in an outpatient setting. Phase II is a randomized clinical trial evaluating prazosin versus placebo for 12 weeks in a double-blind, controlled fashion in an outpatient setting. The treatment will last for 12 weeks and outcomes will include symptoms of PTSD and alcohol use. In phase III, subjects will again participate in a laboratory session. This phase of the study will be conducted after at least 6 weeks of treatment while patients are on medication (prazosin or placebo).

Hypotheses:

Primary: The investigators hypothesize that prazosin will be more effective than placebo in reducing trauma-related stress reactivity in a laboratory paradigm, particularly anxiety, craving for alcohol, and hormonal response, in individuals with PTSD and AD.

Secondary: The investigators hypothesize that stress reactivity will have a moderating effect on treatment with prazosin, such that individuals with high levels of stress reactivity will have fewer heavy drinking days, a significant reduction in PTSD symptoms, and shorter time to relapse than individuals with low levels of stress reactivity.

DETAILED DESCRIPTION:
Specific Aim: We propose a laboratory study that will examine stress reactivity as a marker for treatment response to prazosin in patients with PTSD and AD.

Background: Increasing evidence shows that PTSD and AD are both associated with abnormalities in stress reactivity. In PTSD, the increase in hormonal response and subjective increases in affective symptoms provide evidence for abnormalities in stress reactivity. In AD, significant increases in craving after stressful stimuli and alcohol cues point to abnormalities in stress response. There is increasing evidence that these laboratory paradigms are clinically relevant and may be useful in predicting treatment outcomes in patients with substance use disorders. Stress induced craving has been used as a marker for relapse. Individuals with greater stress reactivity have a shorter time to relapse to their preferred substance than individuals with lesser stress reactivity.

Attenuation of trauma-related distress may be effective in reducing both craving and negative affect in individuals with PTSD and AD. In a very elegant study, Coffey and his colleagues (Coffey et al, 2006) found that imaginal exposure therapy was more effective than relaxation alone in reducing craving for alcohol after exposure to stressful imagery and alcohol cues. However, it should be noted that interventions such as imaginal exposure therapy target only symptoms of PTSD, have to be administered by highly trained professionals and have to be provided in specialized settings.

We propose a laboratory study that will test whether pharmacotherapy that targets both symptoms of PTSD and AD can attenuate the stress response, and how the attenuation of stress response will affect relapse and outcome.

Method: This study is designed as an accompaniment to an already funded study by the DOD - a 12-week treatment trial with prazosin for patients with PTSD and AD. The current proposal will augment the findings from the treatment study and identify for which patients prazosin may be effective. It is important to note that this study is very different from the PTSD Coop study in that study EXCLUDES individuals with alcohol dependence. The DOD study and this companion study will provide answers relevant to alcohol use, alcohol relapse and drinking outcomes.

The study design will consist of III phases. In phase I, all subjects will participate in three laboratory sessions to determine their reactivity to stress. Stress reactivity will be measured using: traumatic experiences, stressful non-trauma experiences and neutral experiences, presented randomly. Laboratory sessions will be conducted in an inpatient setting. Phase II is a randomized clinical trial evaluating prazosin versus placebo for 12 weeks in a double-blind, controlled fashion in an outpatient setting. The treatment will last for 12 weeks and outcomes will include symptoms of PTSD and alcohol use. In phase III, subjects will again be admitted to an inpatient unit. This phase of the study will be conducted during the 12th and final week on medication while participants are still receiving prazosin or placebo.

Hypotheses: Primary: We hypothesize that prazosin will be more effective than placebo in reducing trauma-related stress reactivity in a laboratory paradigm, particularly anxiety, craving for alcohol, and hormonal response, in individuals with PTSD and AD. And this will be a marker for treatment response to prazosin in patient with PTSD and AD.

Secondary: We hypothesize that stress reactivity will have a moderating effect on treatment with prazosin, such that individuals with high levels of stress reactivity will have fewer heavy drinking days, a significant reduction in PTSD symptoms, and shorter time to relapse than individuals with low levels of stress reactivity.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients age 21 to 65.
* current diagnosis of DSM-IV PTSD (determined by SCID and CAPS and AD (determine by SCID)).
* participants who drink regularly (determined by TLFB and recorded 90 days prior to the interview), and are not abstinent for more than 2 weeks before participation in the study.
* are not in an active phase of alcohol withdrawal.
* are not at risk for suicide.

Exclusion Criteria:

* current SCID diagnosis of any psychotic disorder.
* history of substance dependence (other than alcohol and nicotine) in the last 30 days.
* current unstable medical condition such as neurological, cardiovascular, endocrine, renal, liver, or thyroid pathology (LFT 5 times normal, abnormal BUN and creatinine, and unmanaged hypertension with BP > 200/120) which in the opinion of the physician would preclude the patient from fully cooperating or be of potential harm during the course of the study.
* taking medication for a psychiatric condition.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2009-01; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Anxiety, craving for alcohol and hormone levels | 12 weeks

SECONDARY OUTCOMES:
treatment efficacy | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ralevski, Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healtcase System, West Haven, Connecticut, United States

REFERENCES:
- [Result] Ralevski E, Southwick S, Jackson E, Jane JS, Russo M, Petrakis I. Trauma- and Stress-Induced Response in Veterans with Alcohol Dependence and Comorbid Post-Traumatic Stress Disorder. Alcohol Clin Exp Res. 2016 Aug;40(8):1752-60. doi: 10.1111/acer.13120. Epub 2016 Jul 1. PMID 27368085